CLINICAL TRIAL: NCT06688851
Title: Patient Specific Implants for the Decompression of Odontogenic Cysts
Brief Title: Patient Specific Implants (PSIs) for the Decompression of Odontogenic Cysts
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Marton Kivovics, associate professor, Semmelweis University
Other Study IDs: SEDCD55
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Odontogenic Cysts; Odontogenic Keratocyst
Keywords: cyst decompression; enucleation; customized implant; Patient Specific Implat (PSI)
MeSH Terms: conditions — Odontogenic Cysts | interventions — Radionuclide Imaging; Cystostomy; Eye Enucleation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Management of the odontogenic cyst using a Patient Specific Implant (PSI): Patients diagnosed with odontogenic cysts are included in this study. Cone Beam Computed Tomography (CBCT) and Intraoral Scans are performed and registered in a software for the design of Patient Specific Implants (PSI). A customized implant is designed and manufactured using Selective Laser Melting (SLM). Under local anesthesia, cystostomy is performed, and the wall of the cyst is sampled for histological diagnosis. The PSI is anchored subperiosteally on the bone using osteosynthesis screws. After a 6-month-long decompression period a CBCT scan is performed to determine whether enucleation of the cyst is feasible. Enucleation of the cyst is performed and the remaining cyst lining is sent for histopathological examination.
  Interventions: Diagnostic Test: Preoperative Cone Beam Computed Tomography (CBCT) scan; Procedure: Cystostomy; Diagnostic Test: Histology to confirm the initial diagnosis; Device: Patient Specific Implant; Procedure: Cyst decompression; Diagnostic Test: CBCT; Procedure: Enucleation; Diagnostic Test: Histology performed on the entire lining of the cyst

INTERVENTIONS:
Diagnostic Test: Preoperative Cone Beam Computed Tomography (CBCT) scan — A CBCT scan is performed before the surgical intervention.
Procedure: Cystostomy — Under local anesthesia, a full-thickness flap is prepared and cystostomy is performed.
Diagnostic Test: Histology to confirm the initial diagnosis — A sample of the cyst lining is sent for histologic diagnosis.
Device: Patient Specific Implant — The PSI is fixed on the surface of the bone using osteosynthesis screws.
Procedure: Cyst decompression — The PSI enables the discharge of the cystic liquid into the oral cavity. The resulting decrease in cystic pressure induces bone healing. Patients are recalled monthly for controls and panoramic X-rays are performed to monitor the decompression.
Diagnostic Test: CBCT — Post-operative CBCT is performed six months after cystostomy to assess whether the cyst volume has been sufficiently reduced for enucleation, minimizing the risk of damage to anatomical landmarks.
Procedure: Enucleation — Under local anesthesia a full-thickness flap is raised and the PSI is removed by unscrewing the osteosynthesis screws. The wall of the cyst is completely enucleated and the flap is sutured.
Diagnostic Test: Histology performed on the entire lining of the cyst — The residual cyst wall is sent for histopathologic examination.

SUMMARY:
This study aims to assess the feasibility of the decompression of odontogenic cysts using Patient Specific Implants anchored subperiosteally using osteosynthesis screws.

DETAILED DESCRIPTION:
Preoperative Imaging and PSIs The digital impression of the dentition or the edentulous jaw is captured using an intraoral scanner and a CBCT scan is performed for each patient enrolled in the study.

Standard Tessellation Language (STL) and Digital Imaging and Communications in Medicine (DICOM) files are imported and registered in the software used for designing the Patient Specific Implants (PSI). The PSI consists of a plate that enables the fixation of the appliance subperiosteally on the bone using osteosynthesis screws and a tube allowing the continuous discharge of the cystic liquid into the oral cavity. The decreased pressure within the cyst enables bone regeneration during the decompression period.

The PSI is produced using Selective Laser Melting (SLM) technology with Titanium. Before the surgical procedure, the PSI undergoes disinfection and sterilization.

Surgical Interventions Under local anesthesia, a full-thickness flap is prepared and cystostomy is performed. A sample of the cyst lining is sent for histological diagnosis. The PSI is fixed on the surface of the bone using osteosynthesis screws. The flap is sutured around the tube of the PSI. After one week the sutures are removed.

Patients are recalled monthly for controls and panoramic X-rays are performed to monitor the decompression.

A post-operative CBCT scan is conducted six months after cystostomy to assess whether the cyst volume has sufficiently decreased for enucleation to be performed with minimal risk of damaging anatomical landmarks.

Under local anesthesia, a full-thickness flap is raised and the PSI is removed by unscrewing the osteosynthesis screws. The wall of the cyst is completely enucleated and the flap is sutured. The residual cyst lining is sent for histopathologic examination.

Data acquisition The complications are documented in the patient's chart after surgical interventions and during follow-up appointments. The volume of the cyst is measured on the CBCT reconstructions before and after decompression to evaluate the effectiveness of the approach described.

ELIGIBILITY:
Inclusion Criteria:

-Patients of the Department of Public Dental Health, Semmelweis University, presenting with odontogenic cysts of the jaws that involve anatomical landmarks are included in the study.

Exclusion Criteria:

* Patients who have uncontrolled major systemic diseases as classified by the American Society of Anesthesiologists (ASA grades III-IV)
* Cancer of the oral cavity
* History of irradiation therapy in the head and neck region within the previous five years,
* History of uncontrolled psychiatric disorders,
* Unwillingness to return for follow-up appointments.
* Patients on medications interfering with bone metabolism, including steroid therapy and antiresorptive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Department of Public Dental Health, Semmelweis University, presenting with odontogenic cysts of the jaws.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Success of the treatment of the odontogenic cyst by the approach described | Decompression may take at least 6 months up to 18 months and lasts until the enucleation may be carried out with minimal risk of complicatios to anatomical landmarks included in the cyst.
  The odontogenic cyst is resolved clinically and radiologically by bony healing
Recurrence | One year after enucleation
  During follow up recurrence of the odontogenic cyst is observed
Intra- and postoperative complications associated with surgery | through study completion, an average of 1 years
  Number of cases where bleeding, damage to neighboring teeth, roots, and anatomical structures, nerve damage, antro-oral communication or fistula, antro-nasal communication or fistula, inflammation is observed during follow up.

SECONDARY OUTCOMES:
Volumetric changes | 6 months to 18 months. The timeframe of decompression.
  Volumetric changes of the cyst cavity during decompression.

CONTACTS AND LOCATIONS:
Overall Officials: Márton Kivovics, Doctor of Dental Medicine, Principal Investigator — Department of Public Dental Health, Semmelweis University
Locations (1):
- Department of Public Dental Health, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) that underlie the results after de-identification.
Supporting Information: Study Protocol
Time Frame: 1 year following the end date
Access Criteria: Immediately following publication. No end date.